CLINICAL TRIAL: NCT07333729
Title: Evaluation of the Impact of Spinal Anesthesia on the Fetal Autonomic Nervous System During an Elective Caesarean Delivery
Brief Title: Effects of Spinal Anesthesia on the Fetal Autonomic Nervous System
Acronym: RACHISNA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024_0479
Record Dates: First submitted 2025-11-24; First posted 2026-01-12 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Obstetrics: Elective Caesarean Delivery
Keywords: Autonomic nervous system; Spinal anesthesia; Hypotension; Fetal heart rate; TOCONAUTE
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TOCONAUTE + ANI RELECTURE (Experimental)
  Interventions: Device: Recording of fetal and maternal heart rate

INTERVENTIONS:
Device: Recording of fetal and maternal heart rate — This study will be conducted in the maternity ward of the Jeanne de Flandre Maternity, Lille University Hospital, specifically in the operating room for cesarean delivery. The TOCONAUTE device will be placed on the mother's abdomen to record fetal heart rate. Recordings will be analyzed retrospectively using the ANI RELECTURE software to calculate the Fetal Stress Index (FSI). Participants will also be connected to the Analgesia Nociception Index (ANI) monitor and the ClearSight system to collect maternal cardiac output, heart-rate variability (HRV) indices, and continuous blood-pressure data. For each participant, the TOCONAUTE will remain in place on the abdomen for 12 minutes after intrathecal injection. These procedures will not interfere with the standard clinical care provided to the pregnant woman.

SUMMARY:
Elective cesarean deliveries account for over 10% of births in France and are often scheduled around 39 weeks of gestation. When feasible, spinal anesthesia is considered the gold standard in such a clinical situation. However, a well-known complication is maternal hypotension, which may lead to placental hypoperfusion and fetal acidosis. Heart rate variability (HRV) markers reflect autonomic nervous system (ANS) activity, which plays a key role in maintaining fetal homeostasis.

The Lille University Hospital has developed a technology to assess parasympathetic activity through HRV analysis. This technology has been adapted to obtain an HRV markers specific of the fetal autonomic nervous system assessment: the Fetal Stress Index (FSI). Preclinical studies have shown that FSI correlates with parasympathetic fluctuations and fetal acidosis.

This pilot study aims to evaluate the impact of spinal anesthesia on fetal ANS activity during elective cesarean delivery using a continuous beat-to-beat fetal heart rate recording device: the TOCONAUTE device. FSI will be retrospectively computed to assess fetal autonomic response. Maternal ANS activity will also be monitored using the Analgesia Nociception Index (ANI). A secondary objective is to explore the predictive value of ANI and FSI for maternal hypotension or fetal hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman scheduled for elective cesarean delivery
* Age: over 18 and under 45 years
* Gestational age ≥ 37 weeks of amenorrhea
* Singleton pregnancy
* Proficient in the French language
* Participant has provided written informed consent to take part in the study
* Affiliated with a national health insurance scheme

Exclusion Criteria:

* Requirement for general anesthesia or combined epidural-spinal analgesia
* Fetal malformation
* Intrauterine fetal demise
* Maternal and/or fetal cardiac rhythm disorders
* History of heart transplantation
* Open wound in an area covered or enclosed by one of the study devices
* Risk of viral or infectious contamination of any component of the device
* Hospitalization for medical termination of pregnancy
* Sensory disorders resulting in lack of pain perception on the skin
* Ongoing treatment that may alter autonomic nervous system activity (e.g., beta-blockers, anticholinergics, atropine)
* Participant with an implanted medical device (e.g., pacemaker)
* Known allergy to any component of the devices: polyamide, polyester, elastane, silver, or other synthetic materials
* Participant whose anatomical area intended for ClearSight sensor placement is insufficient to allow proper application
* Concurrent participation in another interventional research study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2026-12-17 (Estimated)

PRIMARY OUTCOMES:
To assess the impact of spinal anesthesia on fetal autonomic nervous system activity during elective cesarean delivery. | At 12 minutes after intrathecal injection
  Rate of Fetal Stress Index (FSI) compared with the pre-anesthesia baseline, computed from continuous fetal heart-rate recordings acquired with the TOCONAUTE device.

SECONDARY OUTCOMES:
To assess the impact of spinal anesthesia on fetal autonomic nervous system activity at intermediate time points during elective cesarean delivery. | At placement, at injection, 1 min, 3 min, 6 min and 9 min during elective cesarean delivery.
  Rate of Fetal Stress Index (FSI) at multiple intermediate time points after intrathecal injection (at placement, at injection (T0) and at T+1, T+3, T+6, and T+9 minutes) compared with the pre-anesthesia baseline, computed from continuous fetal heart-rate recordings acquired with the TOCONAUTE device.
To evaluate the evolution of maternal blood pressure following spinal anesthesia placement, up to 12 minutes after injection. | At intrathecal injection (T0) and at T+1, T+3, T+6, T+9, and T+12 minutes,
  Change from baseline in ClearSight® (Edwards Lifesciences®) monitoring parameters (systolic arterial pressure (SAP), mean arterial pressure (MAP) measured at intrathecal injection (T0) and at T+1, T+3, T+6, T+9, and T+12 minutes, relative to the pre-spinal anesthesia baseline.
To evaluate the evolution of cardiac output following spinal anesthesia | At intrathecal injection (T0) and at T+1, T+3, T+6, T+9, and T+12 minutes
  Change from baseline in ClearSight® (Edwards Lifesciences®) monitoring parameter: cardiac index (CI) measured relative to the pre-spinal anesthesia baseline.
To evaluate the evolution of cardiac output following spinal anesthesia | At intrathecal injection (T0) and at T+1, T+3, T+6, T+9, and T+12 minutes
  Change from baseline in ClearSight® (Edwards Lifesciences®) monitoring parameter: Hypotension Prediction Index (HPI) measured relative to the pre-spinal anesthesia baseline.
Change in ANI measurements measured at placement, at intrathecal injection (T0) and at T+1, T+3, T+6, T+9, and T+12 minutes, relative to the pre-spinal anesthesia baseline, measured by ANI monitor medical device. | At placement, at intrathecal injection (T0) and at T+1, T+3, T+6, T+9, and T+12 minutes
  Change in ANI measurements measured relative to the pre-spinal anesthesia baseline.
To compare fetal and maternal heart rate variability markers measured during the 12 minutes following spinal anesthesia placement, according to the maternal hypotension status. | At placement, at intrathecal injection (T0) and at T+1, +3, +6, +9, and +12 minutes
  Rate of FSI (Fetal Stress Index) and HPI (Hypotension Prediction Index) measured at placement, at intrathecal injection (T0) and at T+1, +3, +6, +9, and +12 minutes.
To compare fetal and maternal cardiac output values measured during the 12 minutes following spinal anesthesia placement, according to the maternal hypotension status. | At placement, at intrathecal injection (T0) and at T+1, +3, +6, +9, and +12 minutes
  Rate of FSI and ANI measured at placement, at intrathecal injection (T0) and at T+1, +3, +6, +9, and +12 minutes.
To compare fetal and maternal heart rate variability markers measured during the 12 minutes following spinal anesthesia placement, according to the neonatal acidosis status. | At placement, at intrathecal injection (T0) and at T+1, +3, +6, +9, and +12 minutes
  Rate of FSI and HPI measured at placement, at intrathecal injection (T0) and at T+1, +3, +6, +9, and +12 minutes, with analyses stratified by the presence or absence of neonatal acidosis (defined as umbilical arterial pH < 7.20 at birth).
To compare fetal and maternal cardiac output values measured during the 12 minutes following spinal anesthesia placement, according to the neonatal acidosis status. | At placement, at intrathecal injection (T0) and at T+1, +3, +6, +9, and +12 minutes
  Rate of FSI and ANI measured at placement, at intrathecal injection (T0) and at T+1, +3, +6, +9, and +12 minutes, with analyses stratified by the presence or absence of neonatal acidosis (defined as umbilical arterial pH < 7.20 at birth).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No